CLINICAL TRIAL: NCT06847607
Title: A Multicenter Prospective Study of Iptacopan in the Treatment of Refractory/Relapsed Autoimmune Hemolytic Anemia (AIHA)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bing Han (Other)
Responsible Party: Sponsor-Investigator, Bing Han, chief physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIHA-Iptacopan
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: AIHA - Warm Autoimmune Hemolytic Anemia; AIHA - Cold Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iptacopan-AIHA (Experimental): Iptacopan-AIHA
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Iptacopan

SUMMARY:
To evaluate the efficacy and safety of ipecopam in the treatment of refractory/relapsed AIHA.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed an informed consent form (ICF);
2. Males or females aged 18 or older;
3. Physical status score [Eastern Cooperative Oncology Group (ECOG) score] ≤2;
4. Confirmed diagnosis of primary AIHA or secondary autoimmune disease (except rheumatoid arthritis and systemic lupus erythematosus) with underlying disease in a stable state;
5. Poor response to at least previous glucocorticoid therapy, including ineffective (defined as failure to achieve stabilization of Hb levels at 100 g/L or erythrocyte hematocrit <30% despite at least 4 weeks of treatment with previously recommended doses), or glucocorticoid-dependent (defined as maintenance of equal doses of prednisone exceeding 15 mg/d), or relapsed (defined as treatment that is effective and then again has an Hb of <100 g/L or an erythrocyte hematocrit of <30%), or otherwise contraindicated. 30%), or otherwise contraindicated or intolerant to glucocorticoid therapy;
6. Hemoglobin (Hb) <100 g/L before drug administration;
7. Positive direct anti-human globulin test (DAT) (IgA, IgM or IgG+, with or without C3+).
8. Combination of one anti-AIHA therapy [glucocorticoids only (≤15 mg prednisone equivalent), immunosuppressants (azathioprine, cyclosporine, and merti-macrolide only)] is permitted in this study, provided that the dose has been stable for at least 28 days prior to enrollment;
9. Laboratory tests meet the following criteria (no treatment for the abnormality of the index within 2 weeks prior to blood collection, or no long-acting G-CSF treatment within 2 weeks)

   1. Neutrophil count >1.5×109/L and platelet >30×109/L;
   2. ALT and AST ≤ 2 × ULN;
   3. Serum creatinine concentration ≤ 2 × ULN and creatinine clearance ≥ 50mL/min;
10. No active infection; no pregnancy or lactation;
11. cAIHA patients presenting with skin cyanosis and thrombosis;
12. Written evidence of Neisseria meningitidis and Streptococcus pneumoniae vaccinations within 2 years or, if none, antibiotic prophylaxis until 2 weeks after completion of vaccination.

Exclusion Criteria:

1. Presence of secondary AIHA outside the inclusion criteria;
2. Hb <100 g/L due to non-AIHA factors; and
3. Infections requiring systemic therapy;
4. Those with a past history of malignancy (except cured basal cell carcinoma of the skin or cervical carcinoma in situ);
5. With history of vital organ transplantation or hematopoietic stem cell/bone marrow transplantation;
6. Those who have undergone splenectomy within 24 weeks prior to enrollment;
7. Those who have had major surgery within four weeks prior to enrollment or who require major elective surgery during the study period;
8. History of severe cardiovascular disease [e.g., class III/IV congestive heart failure, arrhythmia or angina requiring medication, unstable angina, coronary stenting, angioplasty or coronary artery bypass grafting, or corrected Q-T interval (QTcF) ≥ 90 mmHg]
9. Patients with medically uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg); or comorbid portal hypertension;
10. Patients with severe gastrointestinal disorders such as dysphagia, active gastric ulcers, etc., who are unable to take drugs orally or have impaired absorption of oral drugs;
11. Human immunodeficiency virus (HIV) infection
12. Uncontrolled or active HBV infection [Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) positive patients, need to confirm Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) positive]; or Hepatitis C [patients with Hepatitis C Virus Ribonucleic Acid (HCV RNA) positive patients]; or cirrhosis of the liver;
13. Those who had received herbal treatment within one week prior to enrollment that interfered with the assessment of efficacy;
14. Patients with severe psychological or psychiatric abnormalities;
15. Alcohol or drug abusers;
16. Female patients who are pregnant or breastfeeding;
17. Patients who, in the opinion of the investigator, are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
OR | 3 months
  Overall response rate
CR | 6 months
  complete response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Bing Han, Beijing, China

IPD SHARING:
Plan to Share IPD: No